CLINICAL TRIAL: NCT01510353
Title: Effect of a Real Time Radiation Monitoring Device on Radiation Exposure During Cardiac Catheterization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-097
Record Dates: First submitted 2012-01-09; First posted 2012-01-16 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Radiation Monitoring; Radiation Protection

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Use of a radiation monitoring device (Experimental): Use of a radiation monitoring device that provides real-time auditory feedback on radiation exposure during cardiac catheterization
  Interventions: Device: Radiation monitoring device
- No use of radiation monitoring device (No Intervention): No use of a radiation monitoring device that provides real-time auditory feedback on radiation exposure during cardiac catheterization

INTERVENTIONS:
Device: Radiation monitoring device — Radiation monitoring device (Bleeper Sv, Vertec Scientific Ltd, Berkshire, UK) that provides real-time auditory feedback on radiation exposure during cardiac catheterization
  Arms: Use of a radiation monitoring device

SUMMARY:
The purpose of this study is to examine the impact of using a real time radiation exposure monitoring device on the patient and operator radiation exposure during cardiac catheterization. The hypothesis of the study is that use of a real time radiation exposure monitoring device during cardiac catheterization will decrease both patient and operator radiation exposure compared to no use of the monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically-indicated cardiac catheterization

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Radiation exposure of the operator | radiation exposure will be measured for the duration of the catheterization procedure, an expected average of one hour
  Radiation exposure of the operator (measured in mrem by the real time monitoring device)

SECONDARY OUTCOMES:
Radiation exposure of the patient | radiation exposure will be measured for the duration of the catheterization procedure, an expected average of one hour
  Radiation exposure of the patient, as measured by the X-ray machine using (a) air kerma dose, (b) dose area product, (c) fluoroscopy and cineangiography time

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S. Brilakis, MD, PhD, Study Chair — North Texas Veterans Healthcare System; Subhash Banerjee, MD, Study Director — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

REFERENCES:
- [Derived] Christopoulos G, Papayannis AC, Alomar M, Kotsia A, Michael TT, Rangan BV, Roesle M, Shorrock D, Makke L, Layne R, Grabarkewitz R, Haagen D, Maragkoudakis S, Mohammad A, Sarode K, Cipher DJ, Chambers CE, Banerjee S, Brilakis ES. Effect of a real-time radiation monitoring device on operator radiation exposure during cardiac catheterization: the radiation reduction during cardiac catheterization using real-time monitoring study. Circ Cardiovasc Interv. 2014 Dec;7(6):744-50. doi: 10.1161/CIRCINTERVENTIONS.114.001974. Epub 2014 Nov 25. PMID 25423958